CLINICAL TRIAL: NCT00518154
Title: Pilot Study of an ACh-E Inhibitor Upon Immune Activation Markers in HIV-1 Infected Patients Receiving Highly Active Antiretroviral Therapy (HAART) Showing an Incomplete Immune Response.
Brief Title: Pilot Study of Pyridostigmine Upon Immune Activation in HIV-1 Patients Who Have an Inadequate Immune Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Sergio I. Valdés-Ferrer, MD, PhD, Investigator, Depatment of Infectious Diseases, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ref. 1663
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: HIV Infections
Keywords: AIDS; Immunological non-responders; Neuroimmune modulation; Pyridostigmine; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Patients will be taking oral Pyridostigmine 30mg tid, as well as their usual antiretroviral treatment
  Interventions: Drug: Pyridostigmine tablets

INTERVENTIONS:
Drug: Pyridostigmine tablets — Patients will take 30mg tid PO for 12 weeks
  Other Names: Mestinon

SUMMARY:
The purpose of this study is to determine whether the addition of Pyridostigmine to Highly Active Antiretroviral Therapy (HAART) increases the number of CD4+ T-cells in discordant patients in which viral load diminishes, but T-cell levels remain low after the initiation of treatment.

DETAILED DESCRIPTION:
In HIV-1 infected patients, HAART suppresses viral replication, reflected by a reduced viral load, and a recovery in the frequency of CD4+ T-cells. The latter is associated with a reduced risk for developing opportunistic infectious diseases, and death. T-cell recovery, however, is highly variable within individuals, suggesting that virological eradication is but one factor of it.

A phenomenon known as Immune Discordance has been well known. It reflects a subpopulation -as high as 30% of patients- in whom there is an adequate suppression of viral replication, but CD4+ cell levels rise modestly (below safety levels). In this setting, patients remain susceptible to develop opportunistic infections, have disease progression, and die. Various mechanisms have been proposed, but one common factor is enhanced CD4+-cell activation, leading to cell dysfunction and apoptosis.

It is known that an inflammatory response is able to activate the anti-inflammatory cholinergic pathway, in which acetylcholine (ACh) is released and in turn activates nicotinic receptors in macrophages. The result is a diminished synthesis of inflammatory cytokines such as TNF-α, and IL-1. We have recently shown in an ex-vivo, proof-of-concept study carried in HIV-infected subjects in early phases of the infection (not requiring specific treatment) that Pyridostigmine diminishes CD4+-cell activation and an increase in the subpopulation of regulatory T-cells (T-reg).

Pyridostigmine, an ACh-esterase inhibitor, has been shown to be safe in other populations, including healthy Gulf War military personnel, and patients with Myasthenia Gravis. Its hypothetical effect is by reducing the degrading rate of the naturally occurring ACh (released by the vagus nerve) by the enzyme ACh-esterase. This in turn enhances its coupling to nicotinic receptors in macrophages that, according to our previous study (unpublished data), improves the T-cell milieu, diminishes T-cell activation (a well known trigger for apoptosis), and enhances T-reg proliferation.

The purpose of this study is to determine whether the addition of Pyridostigmine to Highly Active Antiretroviral Therapy (HAART) increases the number of CD4+ T-cells in discordant patients in which viral load diminishes, but T-cell levels remain low after the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected subjects 18 years of age or older
* Receiving HAART for at least two years
* At least a viral load determination per year since HAART initiation, all undetectable
* Patient's status is Immunological Non Responder (InR), that is, his or her viral load is reduced, but CD4+ cell count has not raised accordingly
* Current viral load: undetectable
* Patient agrees and signs informed consent

Exclusion Criteria:

* Concomitant active infectious or neoplastic disease
* History of new AIDS-defining events during HAART
* Pregnancy or breast-feeding
* Patients who have been subjects of an investigational agent, chemotherapy or radiotherapy within the previous 28 days
* Subjects requiring treatment for Tuberculosis
* Subjects unable to follow, or comply with the protocol interventions
* Subjects receiving immunosuppressive treatment, including corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sierra-Madero, MD, Study Chair — Dept. of Infectious Diseases, INNSZ; Jorge Alcocer-Varela, MD, Study Director — Dept. of Immunology, INNSZ; Sergio I Valdés-Ferrer, MD, PhD, Principal Investigator — Dept. of Neurology, INNSZ
Locations (2):
- Mexico (2):
  - Sergio I. Valdés-Ferrer, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Tlalpan, Mexico City

REFERENCES:
- [Derived] Valdes-Ferrer SI, Crispin JC, Belaunzaran-Zamudio PF, Rodriguez-Osorio CA, Cacho-Diaz B, Alcocer-Varela J, Cantu-Brito C, Sierra-Madero J. Add-on Pyridostigmine Enhances CD4+ T-Cell Recovery in HIV-1-Infected Immunological Non-Responders: A Proof-of-Concept Study. Front Immunol. 2017 Oct 18;8:1301. doi: 10.3389/fimmu.2017.01301. eCollection 2017. PMID 29093707
- See also: Institute's web page — http://www.innsz.mx

RESULTS

PARTICIPANT FLOW:
Groups:
- Pyridostigmine: Patients will be taking oral Pyridostigmine 30mg tid, as well as their usual antiretroviral treatment. The study is open-label, proof-of-concept.
  Pyridostigmine tablets: Patients will take 30mg tid PO for 12 weeks
Period: Overall Study
Arm/Group | Pyridostigmine
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Change in Circulating CD4+ T-cell Count (Baseline vs. 16 Weeks: Participants will receive pyridostigmine 30mg three times per day for a period of 16 weeks. Pyridostigmine will be in addition (add-on) to their usual antiretroviral treatment schedule.
Arm/Group | Change in Circulating CD4+ T-cell Count (Baseline vs. 16 Weeks
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 7

OUTCOME MEASURES:

1. Primary Outcome: CD4+ Cell Count Change Between Basal and Week 16 of Additive Treatment
Description: Change in total CD4+ T-cell number from baseline to addition of pyridostigmine
Time Frame: 16 weeks after initiation of pyridostigmine
Population: Change in total CD4+ T-cell counts
Measure: Mean (Standard Deviation); unit: CD4+ T-cell count/uL
Arm/Group | Pyridostigmine
Number analyzed (Participants) | 7
CD4+ T-cell count/uL | 153.2 (43.1)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: We will use the standard definition of adverse event: "Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research."
Groups:
- Pyridostigmine: Patients will be taking oral Pyridostigmine 30mg tid, as well as their usual antiretroviral treatment
  Pyridostigmine tablets: Patients will take 30mg tid PO for 12 weeks
Arm/Group | Pyridostigmine
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No